CLINICAL TRIAL: NCT01549444
Title: Renin and Aldosterone Levels in the Preterm Neonate At Risk for Hypertension (RENAL HIT Study)
Brief Title: Renin and Aldosterone Levels in the Preterm Neonate At Risk for Hypertension
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Australian National University (Other)
Responsible Party: Sponsor
Other Study IDs: Renin HIT study-01; NCT01545895 (obsolete NCT alias)
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension; Diabetes; Infants Small for Gestational Age
Keywords: renin; aldosterone; neonate
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for Renin and Alsosterone, to be discarded when study is complete.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Babies of mothers that have diabetes and/or hypertension and babies that are small for dates
  Interventions: Other: presence of maternal risk factor for hypertension
- Group 2: Babies born to mothers without diabetes and/or hypertension and babies that are correct size for gestational age

INTERVENTIONS:
Other: presence of maternal risk factor for hypertension
  Groups: Group 1

SUMMARY:
The purpose of this study is to find out if mothers with high blood pressure (Hypertension) and/or diabetes have babies with high levels of different substances (that help to regulate blood pressure, called Renin and Aldosterone) in their blood. The investigators are also trying to determine if these babies have higher blood pressure than those babies born to mothers without high blood pressure or diabetes, during the first year of life.

The investigators will measure your baby's blood pressure once a day for the first 4 days, at 1 week of age, and then once per week until your baby is discharged. The investigators will also measure the blood pressure after discharge at 4 and 10 months of age, either on the day of your baby's follow-up appointment in the Neonatal Follow-up Clinic or at a visit to our Outpatient Nephrology Clinic, both at CHEO.

DETAILED DESCRIPTION:
We will compare two groups of babies born between 26+0 and 34+0 weeks gestation.Group 1 is the babies born to mothers with diabetes and/or high blood pressure, and babies that are small for dates. Group 2 are babies that are 26 to 34 weeks of age, that are born to mothers without these problems.

In the study we will measure the baby's blood pressure once a day for the first 4 days, at 1 week of age, and then once per week until the baby is discharged. We will also measure the blood pressure after discharge at 4 and 10 months of age, either on the day of your baby's follow-up appointment in the Neonatal Follow-up Clinic or at a visit to our Outpatient Nephrology Clinic, both at CHEO.

As blood tests will be done. A small amount of extra blood, 0.75ml - 1.5 ml (about 1/6 -1/3 of a teaspoon, or approximately 1 ml) will be collected for measurement of the blood substances we are studying will be collected when the baby has their regular non-study blood work.

This will be done within six hours of birth and then again at 2-3 weeks of life.

ELIGIBILITY:
Inclusion Criteria:

1. Infants < 6 hours of age who require NICU admission
2. Infants 26+0 to 34+0 weeks gestation.

Exclusion Criteria:

* Immediate Exclusion from Enrollment

  1. Maternal treatment with drugs known to be teratogenic and cause nephrotoxicity in the fetus (i.e. ACE-Inhibitor).
  2. Infants with known congenital anomalies and/or renal anomalies.
  3. Infants with known chromosomal anomalies.
  4. Infants with severe asphyxia defined as cord pH < 7.0, 5 min Apgar < 3, and urine positive for blood.
  5. Infants with a known or suspected blood loss at birth (ie: uterine rupture, placental abruption, bleeding placenta previa, or post-natal blood loss in the delivery room).
  6. Infants who will not receive follow-up care in Ottawa upon discharge from the NICU (ie: live out of town).

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies born between 26 and 34 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Renin and Aldosterone levels corelated to BP measurements | at birth and at 2-3 weeks of age
  We hypothesize that infants with higher levels of RE and ALDO at birth and in the early neonatal period will have a higher BP during the first year of life.

SECONDARY OUTCOMES:
Blood pressure measurements | in the first month of life, then at 4 and10 months of age
  We hypothesize that premature infants of mothers with hypertension (HT) and/or diabetes, or who are significantly growth restricted will have a higher blood pressure (BP) in the first year of life.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Bariciak, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario